CLINICAL TRIAL: NCT06516497
Title: Use of Motion Sensors in Correction Procedures of Long Bone Deformities in the Pediatric Age Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muhammed Cagatay Engin, ASSOCIATE PROFESSOR, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 536
Record Dates: First submitted 2024-07-13; First posted 2024-07-24 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Angulation Deformity of Long Bone (Disorder); Acquired Deformity of Knee Joint (Disorder)
Keywords: pediatric orthopedics; Deformities; Motion sensor
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group using traditional method in long bone deformity correction (Experimental): 20 people between the ages of 2-18. Pediatric patients with long bone deformities and surgical indications. When correcting the deformity in these patients, the current method in deformity surgery all over the world is roughly corrected and the decision is made according to clinical experience.
  Interventions: Other: Group using traditional method in long bone deformity correction
- Group using computer-aided sensors in long bone deformity correction (Experimental): 20 people between the ages of 2-18. Pediatric patients with long bone deformities and surgical indications. A sensor designed together with engineers will be used to correct the deformity in these patients.
  Interventions: Device: Group using computer-aided sensors in long bone deformity correction

INTERVENTIONS:
Other: Group using traditional method in long bone deformity correction — Osteotomy will be performed from the deformity center after two coring wires are placed in the same plane from the proximal and distal of the determined osteotomy line to the femur or tibia of the patients in the control group with deformity. While the degree of deformity is corrected, the determination will be made after the amount of deformity determined preoperatively is determined visually.
  Arms: Group using traditional method in long bone deformity correction
Device: Group using computer-aided sensors in long bone deformity correction — After 2 wires are placed in the same plane from the proximal and distal parts of the osteotomy line determined on the deformed femur or tibia of patients who underwent general anesthesia during the surgery, motion sensors will be placed on the wires. Osteotomy will be performed on the bone with deformity from the deformity center. When correcting the degree of deformity, the detection will be performed after the correction is achieved by the amount of deformity determined preoperatively.
  Arms: Group using computer-aided sensors in long bone deformity correction

SUMMARY:
Motion sensors will be used in long bone deformity surgery in pediatric patients.

In patients whose deformity status is determined before the surgery, 2 wires will be placed in the same plane from the proximal and distal of the determined osteotomy line to the long bones of the patients who are anesthetized during the surgery and motion sensors will be placed on the wires. Osteotomy will be performed on the bone with deformity from the deformity center. While correcting the degree of deformity, fixation with plate and screws will be performed after the amount of correction determined preoperatively is achieved. Thanks to the sensors and application, it will be determined exactly how many degrees of deformity will be corrected in the case. At the same time, multiplanar and difficult-to-detect deformities will be corrected almost ideally with the help of motion and acceleration sensors. Approximately at the 6th week after the case, deformity correction status will be recorded again with gait analysis and physical examination following the removal of the cast, splint and bone healing. The results will be compared after the traditional method and the method using sensors are performed with an equal number of patients. As a result, it is aimed to clearly correct the deformity quantitatively and shorten the surgical time.

DETAILED DESCRIPTION:
Patients who are between the ages of 2 and 18, who are admitted to Atatürk University Faculty of Medicine Research Hospital, who are considered to have long bone deformities in their lower extremities and who have gait disorders and who have not previously undergone lower extremity surgery, will be included in the study. To determine the degree of preoperative deformity of these patients, a physical examination will be performed after gait analysis and foot advancement angles, hip rotation degrees, thigh foot angles, transmalleolar axis angles and forefoot alignment will be determined and recorded. Following the routine preoperative computerized tomography performed on the patients, long bone alignment disorders, joint incompatibilities (valgus, varus deformities), femoral anteversion, femoral retroversion, tibial torsion angles will be determined quantitatively, and the amount of deformity correction to be performed in the surgery will be determined before the surgery and the quantitative values will be recorded. After two wires are placed in the same plane from the proximal and distal parts of the determined osteotomy line, motion sensors will be placed on the long bones of the anesthetized patients during the surgery. Osteotomy will be performed on the bone with deformity from the deformity center. When correcting the degree of deformity, fixation with plate and screws will be performed after the correction is achieved by the amount of deformity determined preoperatively. (In other countries and in our country, approximate correction is provided without quantitative data. Although the preoperative degree of deformity can be determined quantitatively, surgery is performed by determining the degree of correction intraoperatively by eye decision.) Thanks to the sensors and application, exactly how many degrees of deformity will be corrected will be determined in the case. At the same time, multiplanar and difficult-to-detect deformities will be corrected almost ideally with the help of motion and acceleration sensors. Approximately at the 6th week after the case, deformity correction status will be recorded again with gait analysis and physical examination following the removal of the cast, splint and bone healing.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of long bone deformity
2. Must be between the ages of 2 and 18 when applying for deformity correction.

Exclusion Criteria:

1. Patients or their parents do not accept surgical treatment
2. Not being between the ages of 2 and 18

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
measuring preoperative deformity angles | 2 months
  A preoperative clinical examination will be performed in pediatric orthopedic deformity patients, especially in patients who lean in, lean out, or cannot fully extend their knees. During the clinical examination, measurements will be made with a goniometer or on a computer by taking photographs. For rotational deformities in the transverse plane, the foot advancement angle, femoral internal and external rotation angles, and transmalleolar axis angle will be measured and noted. In patients with extension limitation, the degree of limitation will be measured by goniometer or conventional radiographs. The amount of deformity will be determined exactly and the surgery will be performed.
measuring postoperative deformity angles | 2 months
  The amount of deformity corrected after surgery will be measured and noted by clinical examination and conventional x-rays 2 months later, after the child has recovered.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes